CLINICAL TRIAL: NCT03123003
Title: Bone Age Assessment in Children Using Ultrasound Compared to Wrist X-ray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MeirMc0042-17CTIL
Record Dates: First submitted 2017-03-08; First posted 2017-04-21 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Short Stature; Growth Disorders
Keywords: Bone age,; Height prediction; Growth
MeSH Terms: conditions — Dwarfism; Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SonicBone Ultrasound (Experimental): Assessment of bone age by SonicBone Ultrasound will compared to wrist X-ray assessment
  Interventions: Device: SonicBone Ultrasound; Device: Wrist X-ray

INTERVENTIONS:
Device: SonicBone Ultrasound — Bone age assessment by SonicBone Ultrasound. The patient needs to put his/her wrist in 3 positions.
Device: Wrist X-ray — Bone age assessment by Wrist X-ray

SUMMARY:
Bone age assessment in children is based on the interpretation of hand x-ray scans according to Greulich and Pyle (GP) standard atlas and frequently used for evaluating growth and puberty in children and adolescents.

To address the disadvantage of repeated irradiation, the need for specialized radiation centers, heavy equipment and subjective reading a new device, SonicBone was developed. SonicBone utilizes a quantitative ultrasonographic technology of ultrasonic (US) waves, propagating along a measured bone distance. The aim of the study is to evaluate an ultrasound based device, SonicBone, compared to the current method in children. The investigators will be compared the US assessment to available bone age X-ray that exists in the medical files of the patients. The investigators will not do bone age X-ray scans especially for the current study.

DETAILED DESCRIPTION:
Bone age assessment in children is based on the interpretation of hand x-ray scans according to Greulich and Pyle standard atlas and frequently used for evaluating growth and puberty in children and adolescents.

To address the disadvantage of repeated irradiation, the need for specialized radiation centers, heavy equipment and subjective reading a new device, SonicBone was developed. SonicBone utilizes a quantitative ultrasonographic technology of ultrasonic (US) waves, propagating along a measured bone distance. The aim of the study is to evaluate the ultrasound based device, SonicBone, and to compare it to the current method used in children.

The SonicBone device (Rishon Lezion, Israel) is a small (50cm X 25cm X 25cm), portable, bone sonometer, which measures two parameters:

1. speed of propagation through bone (speed-of-sound, SOS, m/sec) of inaudible high frequency waves of a short ultrasound pulse; and
2. attenuation (ATN; the decay rate) of the sound wave by the bone as a function of the distance it travels between a transmitter probe and a receiver probe15. The hand is measured by: 1- wrist (W), measuring SOS and ATN at the distal radius and ulna secondary ossification centers of the epiphyses; 2-metacarpals (MC), measuring SOS and ATN at the distal metacarpal epiphyses; and 3- phalange (P), measuring SOS and ATN along the bent proximal third phalanx shaft, growth plate and epiphysis. The average of those 3 readings is define as the child's bone age by SonicBone. All ultrasonic examinations will be conducted at the Pediatric Endocrinology Clinic, by a trained technician.

X-ray scans will be evaluated independently by a pediatric endocrinologist according to the GP atlas.

ELIGIBILITY:
Inclusion Criteria:

* Children 3.5-18 years old refered to the endocrine pediatric clinic due to short stature or other growth abnormalities

Exclusion Criteria:

* Children with bone disease
* Children who within the last year took medications which might change bone metabolism or mineralization

Ages: 42 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
bone age | through study completion, an average of 1 year
  Bone age in years

CONTACTS AND LOCATIONS:
Overall Officials: Alon Eliakim, Prof., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No